CLINICAL TRIAL: NCT02952547
Title: A Randomized, Open-label, Oral Dose, Crossover Study to Compare the Safety and Pharmacokinetics Between Co-administration and Fixed Dose Combination of DWC20155 and DWC20156 in Healthy Subjects
Brief Title: Safety and Pharmacokinetics Study of DWC20155 and DWC20156 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1366002
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test / Reference Drug (Experimental): DWJ1366 Tab. followed by co-administration of DWC20155 and DWC20156 Tab.
  Interventions: Drug: Co-administration of DWC20155 and DWC20156; Drug: DWJ1366 Tab.
- Reference / Test Drug (Experimental): Co-administration of DWC20155 and DWC20156 Tab. followed by DWJ1366 Tab.
  Interventions: Drug: Co-administration of DWC20155 and DWC20156; Drug: DWJ1366 Tab.

INTERVENTIONS:
Drug: Co-administration of DWC20155 and DWC20156
Drug: DWJ1366 Tab.

SUMMARY:
The purpose of this study to Compare the safety and pharmacokinetics between co-administration and fixed dose combination of DWC20155 and DWC20156 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.5 and ≤ 27.0 kg/m2.
* No clinically significant findings
* Age 19-55 years at screening

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2016-11-26 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0-24 hours
Area under the plasma concentration versus time curve (AUC) | 0-24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No